CLINICAL TRIAL: NCT00942578
Title: A Phase 2 Trial of Bevacizumab, Lenalidomide, Docetaxel, and Prednisone (ART-P) for Treatment of Metastatic Castrate-Resistant Prostate Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Ravi A. Madan, M.D., Principal Investigator, National Institutes of Health Clinical Center (CC)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 090195; 09-C-0195
Record Dates: First submitted 2009-07-18; First posted 2009-07-21 (Estimated); Results first posted 2018-10-11 (Actual); Last update posted 2018-10-11 (Actual); Status verified 2018-09

CONDITIONS: Metastatic Prostate Cancer
Keywords: Dual Antiangiogenic Combination Therapy for mCRPC; Efficacy and Toxicity Profile; Single Stage Phase 2 With Early Stopping, Run In Phase For Toxicity; Correlative Measurements; Overall Survival Assessment; Metastatic Prostate Cancer; Prostate Cancer
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Bevacizumab; Lenalidomide; Docetaxel; Prednisone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Single Arm - 4 Drug Combination (Experimental): A two dose level escalation of Lenalidomide from 15mg to 20mg to 25mg- standard 3+3 dose escalation approach in combination with docetaxel, Bevacizumab and prednisone.
  Interventions: Drug: Bevacizumab; Drug: Lenalidomide; Drug: Docetaxel; Drug: Prednisone

INTERVENTIONS:
Drug: Bevacizumab — 15 mg/kg cycle 1 day 1, repeated every 21 days
  Other Names: Avastin
Drug: Lenalidomide — Once daily days 1-14 of every 21
  Other Names: Revlimid
Drug: Docetaxel — 75 mg/m^2 intravenous (IV) over 60 minutes on cycle 1 day 1, repeated every 21 days (a 3-week cycle)
  Other Names: Taxotere
Drug: Prednisone — 10 mg orally every day
  Other Names: Deltasone

SUMMARY:
Background:

* Prednisone and docetaxel have been used successfully in treating patients with prostate cancer, either when used alone or in combination with other agents. Researchers believe that these anticancer effects can be increased by giving them in this specific combination.
* A previous study at the National Cancer Institute combined docetaxel and prednisone with bevacizumab and thalidomide. The results of this study were promising; however, most patients in the study required a dose reduction of thalidomide because of its side effects.
* Lenalidomide, a drug similar to thalidomide, may have less severe side effects. Based on previous studies, lenalidomide is well tolerated in patients with solid tumors when used alone or in combination with docetaxel, and it may be a good substitute for thalidomide.

Objectives:

* To determine if lenalidomide is an appropriate and effective substitute for thalidomide in treating prostate cancer.
* To evaluate the safety and effectiveness of bevacizumab, lenalidomide, docetaxel, and prednisone as a prostate cancer treatment, and to study any side effects.

Eligibility:

- Men 18 years of age and older who have been diagnosed with metastatic prostate cancer that has not responded to standard treatment, including surgical removal of the testicles or treatment with androgen (sex-hormone) suppressing drugs.

Design:

* Participants will have a complete medical history and physical examination before beginning the study.
* Patients will be treated with 21-day cycles with a combination of four drugs:
* (1) Docetaxel, which will be given into a vein for 60 minutes on the first day of each 21-day cycle. Patients will take dexamethasone (a steroid agent) before and after taking docetaxel.
* (2) Prednisone, which will be taken by mouth daily.
* (3) Bevacizumab, which will be given through a vein over 30 to 90 minutes on the first day of each 21-day cycle following the infusion of docetaxel.
* (4) Lenalidomide, which will be taken by mouth during the first 2 weeks of each 21-day cycle. The dose of lenalidomide may be adjusted if side effects develop.
* Patients will also receive enoxaparin, a subcutaneous injection administered daily, to prevent blood clots and/or pegfilgrastim, a subcutaneous injection on day 2 of each cycle, to improve white blood cell counts, as directed by researchers.

DETAILED DESCRIPTION:
Background:

The dual antiangiogenic therapy with bevacizumab and thalidomide in combination with docetaxel and prednisone (ATTP) is highly active in patients with metastatic castration resistant prostate cancer (mCRPC), associated with unprecedented results (90% patients had PSA declines of greater than or equal to 50% and 64% ORR in measurable disease).

Most patients in the ATTP trial required dose reduction due to thalidomide toxicities.

Lenalidomide, an analogue of thalidomide, possesses both antiangiogenesis and inhibition of TNF-alpha, but has a favorable toxicity profile. Lenalidomide is well tolerated in patients with solid tumors when used alone or in combination with docetaxel.

To preserve the efficacy of ATTP and to potentially reduce toxicity, lenalidomide may be a good substitute for thalidomide.

Objectives

Primary:

To assess if lenalidomide at its approved dosing schedule can be safely combined with docetaxel, bevacizumab, and prednisone in patients with mCRPC (less than 25% Grade 4 toxicity)

To evaluate the efficacy of the combination

Eligibility:

Patients with progressive mCRPC who have not received any chemotherapy or antiangiogenic therapy for mCRPC

Design:

A single-stage Phase 2 study, with an early stopping rule for excessive toxicity: the goal is to enroll 45 patients at the 25-mg dose level of lenalidomide. However, if 7 in the first 18 or fewer patients receiving lenalidomide at 25 mg develop grade 4 non-hematologic toxicity at anytime during study, no further patients will be enrolled. With respect to the stopping rule, a grade 4 hematologic toxicity will be considered if the episode has lasted for greater than or equal to 5 days. Grade 4 lymphopenia of any duration will not be counted. If less than 7 of the first 18 patients experience the above level of toxicity, accrual will continue until 45 patients have been enrolled at the 25 mg dose level of lenalidomide.

A run-in phase with lenalidomide at 15 mg will be conducted in the first three patients and at 20mg for the next three patients for assessing its tolerability within the combination prior to dosing at 25 mg thereafter.

An expansion cohort of a lower dose of lenalidomide (15 mg) in combination with docetaxel and and Avastin will be conducted to asses if this lower dose of lenalidomide could have similar efficacy with less toxicity.

Treatment Schema of ART-P

Dex -Dexamethasone 8 mg. po 12 hours pre, 3 hours pre, and 1 hour pre infusion of docetaxel (patients who were on prior regimen which included a lower dose of decadron and did not have a reaction do not have to increase their decadron to the 8 mg dose)

Len - Lenalidomide 25 mg po, days 1-14. Lenalidomide 15 mg and 20mg for the proposed run-in phase. Lenalidomide 15 mg for the expansion cohort.

Doc - Docetaxel 75 mg/m2 IV

Bev - Bevacizumab 15 mg/kg IV

Pre - Prednisone 10 mg PO daily throughout cycle

E - Enoxaparin given SQ daily based on weight (see dosing chart in section 4.2)

Peg - Pegfilgrastim 6mg SQ given at least 24 hours after docetaxel administration

Baseline screening evaluations are to be conducted within 15 days prior to protocol enrollment. Baseline scans and x-rays must be performed 4 weeks prior to protocol enrollment. Patients must be evaluated at the NCI clinic each cycle for treatment continuation. Staging scans will be performed after the first 2 cycles of treatment and then every three cycles. All follow-up evaluations can be done on the last week of the prior cycle.

ELIGIBILITY:
* INCLUSION CRITERIA:

Castrate-resistant metastatic adenocarcinoma of the prostate defined as progressive metastatic disease (see below) while on GnRH agonists or post surgical castration. All patients enrolled will be required to have evaluable disease on imaging studies.

Histopathological documentation of prostate cancer confirmed in the NCI Laboratory of Pathology at the National Institutes of Health, the Pathology Department at Walter Reed Medical Center, or the Pathology Department at National Naval Medical Center, prior to starting this study. In addition, patients whose slides are lost or unavailable will be eligible for the study if they provide documentation of prostate cancer and if they meet criteria of clinically progressive prostate cancer as outlined (see below).

Clinically progressive prostate cancer documented prior to entry. Progression must be evidenced and documented by any of the following parameters:

i) Two consecutively rising prostatic specific-antigen (PSA) levels apart of 2 weeks

ii) At least one new lesion on bone scans.

iii) Progressive measurable disease.

Patients must have undergone bilateral surgical castration or must continue on GnRH agonist.

Those patients receiving an anti-androgen agent for at least 6 months and are entering the trial due to a rise in PSA must demonstrate a continued rise in PSA 4 weeks after stopping flutamide and 6 weeks after stopping bicalutamide or nilutamide.

May not have received any chemotherapy or antiangiogenic therapy (including thalidomide, lenalidomide, bevacizumab and its targets receptor inhibitors) for metastatic prostate cancer. (Prior immunotherapy/vaccine, experimental hormonal therapy, radiation and (neo)adjuvant chemotherapy is permitted)

Age greater than or equal to 18 years

Eastern Cooperative Oncology Group (ECOG) performance status less than or equal to 2

Must have adequate organ and marrow function as defined below:

Laboratory Test and Required Value:

* Leukocytes greater than or equal to 3,000/microL
* Absolute neutrophil count greater than or equal to 1,500/ microL
* Platelets greater than or equal to 100,000/ microL
* Total bilirubin less than or equal to 1.5 times the institutional upper limits of normal, or less than or equal to 3 mg/dl in a subject with Gilbert Syndrome
* Aspartate aminotransferase (AST) (serum glutamic oxaloacetic transaminase (SGOT) and alanine aminotransferase (ALT) (serum glutamic pyruvic transaminase (SGPT) less than or equal to 2.5 times the institutional upper limit of normal
* Creatinine less than or equal to 1.5 times the institutional upper limits of normal

OR

-Creatinine clearance greater than or equal to 50 mL/min/1.73 m(2) for patients with creatinine levels above institutional normal.

Recovered from any acute toxicity from surgery or radiotherapy, with minimum 4 weeks from major surgical procedures and 2 weeks from radiotherapy

Must be willing to travel from their home to the National Institutes of Health (NIH) for follow-up visits

Able and willing to follow instructions and conform to protocol.

Patients may have had no other active malignancy within the past 2 years with the exception of non-melanoma skin cancer and superficial bladder carcinoma.

No history of myocardial infarction within the past 6 months, uncontrolled congestive heart failure (CHF) or uncontrolled angina pectoris

Patients must agree to use adequate contraception (abstinence; hormonal or barrier method of birth control) prior to the study, during the study, and at least six months after completion. Males must agree to use a latex condom during sexual contact with females of childbearing potential while participating in the study and for at least six months following, even if a man has undergone a successful vasectomy. All patients must be counseled at a minimum of every 28 days about pregnancy precautions and risks of fetal exposure as indicated in the consent.

Subjects must agree not to share study drug and not donate blood, sperm, or semen. A female of childbearing potential is a sexually mature woman who: 1) has not undergone a hysterectomy or bilateral oophorectomy; or 2) has not been naturally postmenopausal for at least 24 consecutive months (i.e., has had menses at any time in the preceding 24 consecutive months).

Ability to understand and the willingness to sign a written informed consent document.

EXCLUSION CRITERIA:

Present clinical signs or symptoms of current active brain and/or leptomeningeal metastases confirmed by computed tomography (CT) or magnetic resonance imaging (MRI) brain scan. Patients with previously treated brain metastases are allowed to participate in the study.

--Treated brain metastases are defined as having no ongoing requirement for steroids and no evidence of progression or hemorrhage after treatment for at least 3 months, as ascertained by clinical examination and brain imaging (MRI or CT). (Stable dose of anticonvulsants are allowed). Treatment for brain metastases may include whole brain radiotherapy (WBRT), radiosurgery (RS; Gamma Knife, term linear accelerator (LINAC), or equivalent) or a combination as deemed appropriate by the treating physician. Patients with central nervous system (CNS) metastases treated by neurosurgical resection or brain biopsy performed within 3 months prior to Day 1 will be excluded.

Uncontrolled, intercurrent illness including, but not limited to, symptomatic congestive heart failure (American Heart Association (AHA) Class II or worse), unstable angina pectoris

Psychiatric illness/social situations that would limit compliance with study requirements.

Prior history of hypertensive crisis or hypertensive encephalopathy

Proteinuria, as demonstrated by a 24 hour protein of greater than or equal to 2000 mg. Urine protein should be screened by urine analysis. If urine dipstick is greater than 1.0+, then a 24 hour urine collection for total protein will need to be obtained and the level should be less than 2000 mg for patient enrollment.

Serious, non-healing wound, active ulcer, or untreated bone fracture, including tumor-related pathological fracture

Evidence of bleeding diathesis or significant coagulopathy (in the absence of therapeutic anticoagulation)

Human immunodeficiency virus (HIV)-positive patients receiving combination anti-retroviral therapy are excluded from the study because of possible pharmacokinetic interactions with docetaxel, bevacizumab, and/or the combination.

Greater than Grade 2 peripheral neuropathy at baseline

History of allergic reaction to docetaxel, prednisone, lenalidomide and/or bevacizumab or related products.

Patients who are unable to ingest oral medication.

Patients on treatment for venous thromboembolism (VTE).

History of abdominal fistula, gastrointestinal perforation or intra-abdominal abscess within 6 months prior to day 1

Major surgical procedure, open biopsy or significant traumatic injury within 28 days prior to Day 1 therapy

Anticipation of need for major surgical procedures during the course of the study

Core biopsy or other minor surgical procedure, excluding placement of a vascular access device, within 7 days prior to Day 1

Significant vascular disease (e.g., aortic aneurysm, requiring surgical repair, aortic dissection or recent peripheral arterial thrombosis) within 6 months prior to Day 1

Patients with clinically significant cardiovascular disease are excluded

* Inadequately controlled hypertension (HTN) (systolic blood pressure (SBP) greater than 160 mmHg and/or diastolic blood pressure (DBP) greater than 90 mmHg despite antihypertensive medication)
* History of cerebrovascular accident (CVA) within 6 months (see additional requirement for adjuvant protocols), myocardial infarction or unstable angina within 6 months (see additional requirement for adjuvant protocols)
* New York heart association grade II or greater congestive heart failure
* Serious and inadequately controlled cardiac arrhythmia
* Clinically significant vascular disease as stated above

Patients with known hypersensitivity of Chinese hamster ovary cell products or other recombinant human antibodies

Ages: 18 Years to 100 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 63 (Actual)
Dates: Start 2009-07-16 (Actual); Primary Completion 2017-07-31 (Actual); Study Completion 2017-07-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ravi A Madan, M.D., Principal Investigator — National Cancer Institute (NCI)
Locations (1):
- National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Hudes GR, Greenberg R, Krigel RL, Fox S, Scher R, Litwin S, Watts P, Speicher L, Tew K, Comis R. Phase II study of estramustine and vinblastine, two microtubule inhibitors, in hormone-refractory prostate cancer. J Clin Oncol. 1992 Nov;10(11):1754-61. doi: 10.1200/JCO.1992.10.11.1754. PMID 1383436
- [Background] Hudes GR, Nathan F, Khater C, Haas N, Cornfield M, Giantonio B, Greenberg R, Gomella L, Litwin S, Ross E, Roethke S, McAleer C. Phase II trial of 96-hour paclitaxel plus oral estramustine phosphate in metastatic hormone-refractory prostate cancer. J Clin Oncol. 1997 Sep;15(9):3156-63. doi: 10.1200/JCO.1997.15.9.3156. PMID 9294479
- [Background] Pienta KJ, Redman BG, Bandekar R, Strawderman M, Cease K, Esper PS, Naik H, Smith DC. A phase II trial of oral estramustine and oral etoposide in hormone refractory prostate cancer. Urology. 1997 Sep;50(3):401-6; discussion 406-7. doi: 10.1016/S0090-4295(97)00228-8. PMID 9301705

RESULTS

PARTICIPANT FLOW:
Groups:
- 15 mg Dose Lenalidomide; 20 mg Dose Lenalidomide; 25 mg Dose Lenalidomide: A two dose level escalation of Lenalidomide from 15mg to 20mg to 25mg- standard 3+3 dose escalation approach in combination with docetaxel, Bevacizumab and prednisone.
  Bevacizumab: 15 mg/kg cycle 1 day 1, repeated every 21 days
  Lenalidomide: Once daily days 1-14 of every 21
  Docetaxel: 75 mg/m2 IV over 60 minutes on cycle 1 day 1, repeated every 21 days (a 3-week cycle)
  Prednisone: 10 mg orally every day
Period: Dose Escalation Phase
Arm/Group | 15 mg Dose Lenalidomide | 20 mg Dose Lenalidomide | 25 mg Dose Lenalidomide
Started | 3 | 3 | 3
Completed | 3 | 3 | 3
Not Completed | 0 | 0 | 0
Period: Expansion Phase
Arm/Group | 15 mg Dose Lenalidomide | 20 mg Dose Lenalidomide | 25 mg Dose Lenalidomide
Started | 11 | 0 | 43
Completed | 11 | 0 | 43
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- 15 mg Dose Lenalidomide; 20 mg Dose Lenalidomide; 25 mg Dose Lenalidomide: A two dose level escalation of Lenalidomide from 15mg to 20mg to 25mg- standard 3+3 dose escalation approach in combination with docetaxel, Bevacizumab and prednisone.
  Bevacizumab: 15 mg/kg cycle 1 day 1, repeated every 21 days
  Lenalidomide: Once daily days 1-14 of every 21
  Docetaxel: 75 mg/m(2) intravenous (IV) over 60 minutes on cycle 1 day 1, repeated every 21 days (a 3-week cycle)
  Prednisone: 10 mg orally every day
- Total: Total of all reporting groups
Arm/Group | 15 mg Dose Lenalidomide | 20 mg Dose Lenalidomide | 25 mg Dose Lenalidomide | Total
Number analyzed (Participants) | 14 | 3 | 46 | 63
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 8 | 1 | 20 | 29
  >=65 years | 6 | 2 | 26 | 34
Age, Continuous [Mean (Standard Deviation); unit: years] | 64.25 (5.9) | 63.2 (4.95) | 66.07 (8.02) | 64.51 (6.29)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0 | 0
  Male | 14 | 3 | 46 | 63
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 1 | 1
  Not Hispanic or Latino | 14 | 3 | 45 | 62
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 1 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 1 | 1
  Black or African American | 3 | 1 | 14 | 18
  White | 11 | 2 | 30 | 43
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 14 | 3 | 46 | 63
Gleason Score [Count of Participants; unit: Participants] — The Gleason score helps the physician determine whether prostate tissue is normal or different than normal. The Gleason score ranges from 2-10. The lower number means the prostate tissue is normal tissue. The higher number means the prostate tissue is not normal tissue and may be cancer.
  Participants
    ≤6 | 1 | 0 | 3 | 4
    7 | 3 | 1 | 11 | 15
    8 | 4 | 1 | 10 | 15
    9 | 4 | 1 | 18 | 23
    10 | 2 | 0 | 4 | 6
Eastern Cooperative Oncology Group (ECOG) Performance Status [Count of Participants; unit: Participants] — ECOG 0 is defined as normal activity, fully active, able to carry on all pre-disease performance without restriction. ECOG 1 is defined as symptoms, but ambulatory. Restricted in physically strenuous activity, but ambulatory and able to carry out work of a light or sedentary nature (e.g. light housework. ECOG 2 is defined as in bed <50% of the time. Ambulatory and capable of all self-care, but unable to carry out any work activities. Up and about more than 50% of waking hours.
  Participants
    0 | 3 | 0 | 7 | 10
    1 | 11 | 3 | 36 | 50
    2 | 0 | 0 | 3 | 3
Location of Disease [Count of Participants; unit: Participants]
  Bone only | 7 | 1 | 16 | 24
  Bone and lymph nodes | 1 | 2 | 24 | 27
  Bone and visceral (3 hepatic) | 4 | 0 | 3 | 7
  Lymph node alone | 1 | 0 | 2 | 3
  Visceral alone ( bladder and lung) | 1 | 0 | 1 | 2
Alkaline Phosphatase & Lactate Dehydrogenase [Median (Full Range); unit: U/L] — Alkaline phosphatase is a test to assess liver disease and the normal range is 44 to 147 U/L.
  U/L
    Alkaline phosphatase | 124 [53 to 702] | 84 [71 to 121] | 127 [53 to 956] | 125 [53 to 956]
    Lactate dehydrogenase | 209 [174 to 624] | 177 [152 to 193] | 206.5 [127 to 2305] | 206 [127 to 2305]
Prostatic Specific Antigen (PSA) [Median (Full Range); unit: U/L] — Prostatic Specific Antigen (PSA) is a test to assess prostate cancer and the normal values are 4.0 ng/mL and lower.
  U/L | 61.33 [0.48 to 1452] | 61.6 [19.3 to 95.3] | 85.15 [.014 to 3520] | 78.7 [0.14 to 3520]
Hemoglobin [Median (Full Range); unit: g/dL] — Hemoglobin is a protein in the blood that carries oxygen and the normal range for men is 13.5 to 17.5 g/dL.
  g/dL | 12.85 [8.5 to 14.5] | 12.1 [12.0 to 13.2] | 11.9 [7.4 to 14.8] | 12.0 [7.4 to 14.8]

OUTCOME MEASURES:

1. Primary Outcome: Recommended Phase 2 Dose (RP2D)
Description: The RP2D is the dose at which there are no dose-limiting toxicities (defined as a ≥grade 3 hematological toxicity related to lenalidomide).
Time Frame: 3 weeks
Population: Data in this outcome measure is not shown per dose level because the investigator decided to pool the data for analysis since no significant difference was seen at each dose level. Outcome evaluations for cohorts of 3 and 14 patients would carry little scientific value because they are too small.
Measure: Number; unit: mg
Groups:
- Single Arm - 4 Drug Combination: A two dose level escalation of Lenalidomide from 15mg to 20mg to 25mg- standard 3+3 dose escalation approach in combination with docetaxel, Bevacizumab and prednisone.
  Bevacizumab: 15 mg/kg cycle 1 day 1, repeated every 21 days
  Lenalidomide: Once daily days 1-14 of every 21
  Docetaxel: 75 mg/m2 IV over 60 minutes on cycle 1 day 1, repeated every 21 days (a 3-week cycle)
  Prednisone: 10 mg orally every day
Arm/Group | Single Arm - 4 Drug Combination
Number analyzed (Participants) | 63
mg | 25

2. Primary Outcome: Count of Participants With Dose-Limiting Toxicities (DLT)
Description: DLT is defined as a ≥grade 3 non-hematological toxicity related to lenalidomide.
Time Frame: First 28 days of treatment.
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Single Arm - 4 Drug Combination
Number analyzed (Participants) | 63
Participants | 0

3. Primary Outcome: Median Time to Progression (TTP)
Description: TTP is evaluated from the on-study date until the date of progression or last follow-up after progression.
Time Frame: median time of potential follow-up of 47.5 months
Population: as for outcome 1
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Single Arm - 4 Drug Combination
Number analyzed (Participants) | 63
Months | 18.2 [15.2 to 26.1]

4. Secondary Outcome: Median Overall Survival of Patients Studied
Description: OS is evaluated from the on-study date until the date of death or last follow-up.
Time Frame: median time of potential follow-up of 47.5 months
Population: as for outcome 1
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Single Arm - 4 Drug Combination
Number analyzed (Participants) | 63
Months | 24.6 [21.7 to 31.2]

5. Secondary Outcome: Count of Participants With Changes in Circulating Apoptotic Endothelial Cells (CAEC) From Baseline After Drug Administration
Description: The definition of an increase is any increase (any number greater than zero) in the percent CAEC among total peripheral blood mononuclear cells comparing each patient's percent CAEC among total peripheral blood mononuclear cells at baseline to each patient's percent CAEC among total peripheral blood mononuclear cells at cycle 3 day 1. The definition of a decrease is any decrease (any number less than zero) in the percent CAEC among total peripheral blood mononuclear cells comparing each patient's percent CAEC among total peripheral blood mononuclear cells at baseline to each patient's percent CAEC among total peripheral blood mononuclear cells at cycle 3 day 1.
Time Frame: After drug administration, an average of 3 months
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Single Arm - 4 Drug Combination
Number analyzed (Participants) | 63
Participants
  Increase in CAEC after 3 months | 30
  decrease in CAEC after 3 months | 20

6. Secondary Outcome: Changes in the Molecular Markers of Angiogenesis (i.e Serum VEGF) Before and After Administration of Docetaxel, Prednisone,Lenalidomide and Bevacizumab
Description: Serum and urine samples were collected before and after administration of Docetaxel, Prednisone, Lenalidomide and Bevacizumab to measure VEGF levels.
Time Frame: median time of potential follow-up of 47.5 months
Population: This outcome measure was not done because the blood samples collected were insufficient for measuring plasma VEGF.
Arm/Group | Single Arm - 4 Drug Combination
Number analyzed (Participants) | 0

7. Secondary Outcome: Survival Based on Expression of Programmed Cell Death Protein 1 (PD-1) on Cluster of Differentiation 8 (CD8) + T Cells
Description: Expression of PD-1 on CD8 + T cells was evaluated by flow cytometry. High and low expression are based on the median values. Patients with a low expression of PD-1 proteins had better survival than those with a high expression.
Time Frame: median time of potential follow-up of 47.5 months
Measure: Median (95% Confidence Interval); unit: Months
Groups:
- 15 mg Dose Lenalidomide; 20 mg Dose Lenalidomide; 25 mg Dose Lenalidomide: A two dose level escalation of Lenalidomide from 15mg to 20mg to 25mg- standard 3+3 dose escalation approach in combination with docetaxel, Bevacizumab and prednisone.
  Bevacizumab: 15 mg/kg cycle 1 day 1, repeated every 21 days
  Lenalidomide: Once daily days 1-14 of every 21 days
  Docetaxel: 75 mg/m(2) intravenous (IV) over 60 minutes on cycle 1 day 1, repeated every 21 days (a 3-week cycle)
  Prednisone: 10 mg orally every day
Arm/Group | 15 mg Dose Lenalidomide | 20 mg Dose Lenalidomide | 25 mg Dose Lenalidomide
Number analyzed (Participants) | 9 | 3 | 37
Months
  Low expression | 21.4 [14.2 to NA] — Not available based on small numbers. | 17.8 [NA to NA] — Not available based on small numbers. | 28.9 [13.1 to 43.3]
  High expression | 22.4 [18.1 to NA] — Not available based on small numbers. | 26.1 [NA to NA] — Not available based on small numbers. | 14.8 [10.1 to 18.2]

8. Secondary Outcome: Survival Based on Expression of T Cell Immunoglobulin and Mucin Domain (TIM-3) on Cluster of Differentiation 8 (CD8) + T Cells
Description: Expression of TIM-3 on CD8 + T cells was evaluated by flow cytometry.
Time Frame: 46.5 months
Measure: Median (95% Confidence Interval); unit: Months
Groups:
- 15 mg Lenalidomide; 20 mg Lenalidomide; 25 mg Lenalidomide: A two dose level escalation of Lenalidomide from 15mg to 20mg to 25mg- standard 3+3 dose escalation approach in combination with docetaxel, Bevacizumab and prednisone.
  Bevacizumab: 15 mg/kg cycle 1 day 1, repeated every 21 days
  Lenalidomide: Once daily days 1-14 of every 21 days
  Docetaxel: 75 mg/m(2) intravenous (IV) over 60 minutes on cycle 1 day 1, repeated every 21 days (a 3-week cycle)
  Prednisone: 10 mg orally every day
Arm/Group | 15 mg Lenalidomide | 20 mg Lenalidomide | 25 mg Lenalidomide
Number analyzed (Participants) | 1 | 1 | 16
Months
  Low expression | 23.6 [NA to NA] — Not available based on small numbers. | NA [NA to NA] — Not available based on small numbers. | 20.2 [13.1 to 32.0]
  High expression | NA [NA to NA] — Not available based on small numbers. | NA [NA to NA] — Not available based on small numbers. | 12.7 [6.7 to 27.6]

9. Secondary Outcome: Count of Participants With a Radiologic Response
Description: Radiologic response was assessed by the Response Evaluation Criteria in Solid Tumors (RECIST) v1.0 criteria. Complete response is disappearance of all target lesions. Partial response is at least a 30% decrease in the sum of the diameters of target lesions, taking as reference the baseline sum diameters. Progressive disease (PD) is at least a 20% increase in the sum of the diameters of target lesions, taking as reference the smallest sum on study (this includes the baseline sum if that is the smallest on study). Stable disease is neither sufficient shrinkage to qualify for partial response nor sufficient increase to qualify for PD, taking as reference the smallest sum diameters while on study.
Time Frame: median time of potential follow-up of 47.5 months
Measure: Count of Participants; unit: Participants
Arm/Group | 15 mg Lenalidomide | 20 mg Lenalidomide | 25 mg Lenalidomide
Number analyzed (Participants) | 4 | 2 | 23
Participants
  Confirmed radiologic PR | 3 | 2 | 20
  Complete Response | 0 | 2 | 0
  Stable Disease | 1 | 0 | 3

10. Secondary Outcome: Count of Participants With Prostatic Antigen-Specific (PSA) Declines
Description: PSA decline is defined as a ≥50% decline in measurable disease. Measurable lesions are defined as those that can be accurately measured in at least one dimension (longest diameter to be recorded) as ≥20 mm by chest x-ray, as ≥10 mm with computed tomography, or ≥10 mm with calipers by clinical exam.
Time Frame: median time of potential follow-up of 47.5 months
Measure: Count of Participants; unit: Participants
Arm/Group | 15 mg Lenalidomide | 20 mg Lenalidomide | 25 mg Lenalidomide
Number analyzed (Participants) | 13 | 3 | 45
Participants
  Participants with PSA>30% | 13 | 3 | 41
  Participants with PSA>50% | 12 | 3 | 40
  Participants with PSA>90% | 5 | 1 | 27
  Not Evaluable | 1 | 0 | 1

11. Secondary Outcome: Count of Participants With Serious and Non-serious Adverse Events Assessed by the Common Terminology Criteria in Adverse Events (CTCAE v4.0) Who Were Administered the Four-Drug Combination
Description: Here is the count of participants with serious and non-serious adverse events assessed by the Common Terminology Criteria in Adverse Events (CTCAE v4.0). A non-serious adverse event is any untoward medical occurrence. A serious adverse event is an adverse event or suspected adverse reaction that results in death, a life threatening adverse drug experience, hospitalization, disruption of the ability to conduct normal life functions, congenital anomaly/birth defect or important medical events that jeopardize the patient or subject and may require medical or surgical intervention to prevent one of the previous outcomes mentioned.
Time Frame: Date treatment consent signed to date off study, approximately 93 months and 22 days.
Measure: Count of Participants; unit: Participants
Arm/Group | 15 mg Dose Lenalidomide | 20 mg Dose Lenalidomide | 25 mg Dose Lenalidomide
Number analyzed (Participants) | 14 | 3 | 46
Participants | 14 | 3 | 46

ADVERSE EVENTS:
Time Frame: Date treatment consent signed to date off study, approximately 93 months and 22 days.
Arm/Group | 15 mg Dose Lenalidomide | 20 mg Dose Lenalidomide | 25 mg Dose Lenalidomide
All-Cause Mortality (participants affected / at risk) | 1/14 | 0/3 | 2/46
Serious Adverse Events (participants affected / at risk) | 13/14 | 3/3 | 45/46
Other Adverse Events (participants affected / at risk) | 14/14 | 3/3 | 46/46
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 15 mg Dose Lenalidomide (N=14) | 20 mg Dose Lenalidomide (N=3) | 25 mg Dose Lenalidomide (N=46)
Anemia (Blood and lymphatic system disorders) | 2 (2) | 0 (0) | 4 (11)
Blood bilirubin increased (Investigations) | 1 (1) | 0 (0) | 0 (0)
Confusion (Psychiatric disorders) | 1 (1) | 0 (0) | 2 (2)
Death NOS (General disorders) | 1 (1) | 0 (0) | 2 (2)
Dehydration (Metabolism and nutrition disorders) | 1 (1) | 2 (3) | 9 (10)
Delirium (Psychiatric disorders) | 1 (1) | 0 (0) | 2 (2)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 2 (3)
Febrile neutropenia (Blood and lymphatic system disorders) | 2 (3) | 0 (0) | 8 (10)
Heart failure (Cardiac disorders) | 1 (1) | 0 (0) | 1 (1)
Hypotension (Vascular disorders) | 1 (1) | 1 (1) | 2 (3)
Infections and infestations - Other, specify (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) — Infection with Grade 3 or 4 neutrophils (ANC <1.0 x 10e9/L): Colon
Lung infection (Infections and infestations) | 1 (1) | 0 (0) | 7 (8)
Neutrophil count decreased (Investigations) | 3 (4) | 3 (4) | 22 (43)
Palmar-plantar erythrodysesthesia syndrome (Skin and subcutaneous tissue disorders) | 1 (3) | 0 (0) | 0 (0)
Platelet count decreased (Investigations) | 2 (4) | 0 (0) | 3 (3)
Small intestinal perforation (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Syncope (Nervous system disorders) | 2 (2) | 0 (0) | 3 (3)
Transient ischemic attacks (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Ventricular arrhythmia (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Anorectal infection (Infections and infestations) | 0 (0) | 1 (2) | 0 (0)
Fever (General disorders) | 0 (0) | 1 (2) | 1 (1)
Infections and infestations - Other, specify (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) — Infection with Grade 3 or 4 neutrophils (ANC <1.0 x 10e9/L): Blood
Myalgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Paroxysmal atrial tachycardia (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Rectal fistula (Gastrointestinal disorders) | 0 (0) | 1 (1) | 2 (2)
Vomiting (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Acute kidney injury (Renal and urinary disorders) | 0 (0) | 0 (0) | 2 (2)
Atrial fibrillation (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 2 (2)
CPK increased (Investigations) | 0 (0) | 0 (0) | 1 (1)
Chest pain - cardiac (Cardiac disorders) | 0 (0) | 0 (0) | 2 (2)
Chest wall pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (2)
Cholecystitis (Hepatobiliary disorders) | 0 (0) | 0 (0) | 1 (1)
Colitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Colonic perforation (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Creatinine increased (Investigations) | 0 (0) | 0 (0) | 1 (1)
Depression (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1)
Diarrhea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 3 (3)
Duodenal ulcer (Gastrointestinal disorders) | 0 (0) | 0 (0) | 2 (2)
Electrocardiogram QT corrected interval prolonged (Investigations) | 0 (0) | 0 (0) | 1 (1)
Enterocolitis infectious (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Fatigue (General disorders) | 0 (0) | 0 (0) | 1 (1)
Fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 2 (2)
Gastric hemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Gastric ulcer (Gastrointestinal disorders) | 0 (0) | 0 (0) | 2 (2)
Gastrointestinal disorders - Other, Diverticulitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Gastrointestinal pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Hematuria (Renal and urinary disorders) | 0 (0) | 0 (0) | 4 (5)
Hypersomnia (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Hypoalbuminemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1)
Hypokalemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1)
Hyponatremia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1)
Hypophosphatemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (2)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Ileus (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Infections and infestations - Other, Bacteremia (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Infusion related reaction (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Lower gastrointestinal hemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Myocardial infarction (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Myositis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Neoplasms benign, malignant and unspecified (incl cysts and polyps) - Other, specify (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 11 (11) | 3 (3) | 36 (36) — Progressive disease
Non-cardiac chest pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Pain (General disorders) | 0 (0) | 0 (0) | 1 (1)
Peripheral sensory neuropathy (Nervous system disorders) | 0 (0) | 0 (0) | 1 (2)
Peritoneal infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Presyncope (Nervous system disorders) | 0 (0) | 0 (0) | 3 (3)
Productive cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Renal and urinary disorders - Other, urethral stricture (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (2)
Scrotal infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Sepsis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Sinus bradycardia (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Skin infection (Infections and infestations) | 0 (0) | 0 (0) | 3 (3)
Skin ulceration (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Thromboembolic event (Vascular disorders) | 0 (0) | 0 (0) | 1 (1)
Tricuspid valve disease (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Upper gastrointestinal hemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 2 (2)
Upper respiratory infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Urinary retention (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1)
Urinary tract infection (Infections and infestations) | 0 (0) | 0 (0) | 3 (3)
Urinary tract obstruction (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1)
Weight loss (Investigations) | 0 (0) | 0 (0) | 1 (2)
Wheezing (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Wound dehiscence (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Osteonecrosis of jaw (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 3 (3)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 15 mg Dose Lenalidomide (N=14) | 20 mg Dose Lenalidomide (N=3) | 25 mg Dose Lenalidomide (N=46)
Abdominal pain (Gastrointestinal disorders) | 3 (3) | 2 (5) | 14 (21)
Acoustic nerve disorder NOS (Nervous system disorders) | 1 (3) | 0 (0) | 0 (0)
Agitation (Psychiatric disorders) | 1 (1) | 1 (1) | 3 (3)
Alkaline phosphatase increased (Investigations) | 1 (2) | 0 (0) | 1 (2)
Allergic rhinitis (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 1 (1) | 11 (11)
Alopecia (Skin and subcutaneous tissue disorders) | 2 (2) | 2 (2) | 33 (33)
Anemia (Blood and lymphatic system disorders) | 6 (49) | 2 (7) | 24 (73)
Anorexia (Metabolism and nutrition disorders) | 3 (4) | 3 (4) | 23 (27)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (5) | 2 (2)
Back pain (Musculoskeletal and connective tissue disorders) | 3 (5) | 1 (1) | 16 (24)
Bone pain (Musculoskeletal and connective tissue disorders) | 2 (2) | 1 (1) | 9 (10)
Bruising (Injury, poisoning and procedural complications) | 2 (2) | 1 (1) | 21 (21)
Cardiac disorders - Other, Small pericardial effusion, asymptomatic (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Chest pain - cardiac (Cardiac disorders) | 3 (5) | 0 (0) | 0 (0)
Colonic hemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Confusion (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0)
Constipation (Gastrointestinal disorders) | 4 (5) | 1 (1) | 19 (27)
Cough (Respiratory, thoracic and mediastinal disorders) | 3 (4) | 1 (1) | 15 (19)
Creatinine increased (Investigations) | 1 (1) | 1 (1) | 6 (8)
Dehydration (Metabolism and nutrition disorders) | 2 (2) | 3 (4) | 16 (29)
Dental caries (Gastrointestinal disorders) | 1 (1) | 0 (0) | 3 (3)
Depression (Psychiatric disorders) | 1 (1) | 1 (1) | 4 (6)
Diarrhea (Gastrointestinal disorders) | 7 (11) | 3 (8) | 31 (79)
Dizziness (Nervous system disorders) | 2 (2) | 3 (9) | 15 (18)
Dry skin (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1) | 12 (15)
Dysgeusia (Nervous system disorders) | 4 (7) | 2 (5) | 30 (33)
Dyspepsia (Gastrointestinal disorders) | 1 (1) | 1 (2) | 6 (7)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 2 (3) | 3 (5) | 21 (34)
Ear and labyrinth disorders - Other, specify (Ear and labyrinth disorders) | 1 (1) | 0 (0) | 0 (0) — R ear pressure d/t dry cerumen impaction which was removed on 1/22/13
Ear pain (Ear and labyrinth disorders) | 1 (1) | 0 (0) | 2 (2)
Edema limbs (General disorders) | 3 (3) | 3 (5) | 21 (29)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 4 (5) | 1 (1) | 27 (33)
Eye disorders - Other, Shrinkage of tear ducts (Eye disorders) | 1 (1) | 0 (0) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 3 (4) | 0 (0) | 4 (5)
Fatigue (General disorders) | 6 (12) | 3 (5) | 29 (45)
Fecal incontinence (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (1)
Fever (General disorders) | 4 (5) | 3 (10) | 12 (23)
Flu like symptoms (General disorders) | 1 (1) | 2 (2) | 2 (3)
Gastroesophageal reflux disease (Gastrointestinal disorders) | 1 (1) | 0 (0) | 3 (3)
Gastrointestinal disorders - Other, Gastroenteritis (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 1 (1)
Gingival pain (Gastrointestinal disorders) | 1 (1) | 1 (1) | 2 (2)
Gum infection (Infections and infestations) | 4 (7) | 1 (1) | 5 (7)
Headache (Nervous system disorders) | 3 (5) | 3 (4) | 7 (7)
Hematuria (Renal and urinary disorders) | 1 (3) | 0 (0) | 3 (3)
Hoarseness (Respiratory, thoracic and mediastinal disorders) | 1 (2) | 0 (0) | 9 (10)
Hypercalcemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 1 (1)
Hyperglycemia (Metabolism and nutrition disorders) | 2 (8) | 0 (0) | 3 (4)
Hyperkalemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 3 (5)
Hypertension (Vascular disorders) | 5 (6) | 1 (1) | 18 (34)
Hypoalbuminemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 3 (6)
Hypocalcemia (Metabolism and nutrition disorders) | 2 (2) | 0 (0) | 0 (0)
Hypoglossal nerve disorder (Nervous system disorders) | 1 (1) | 0 (0) | 1 (1)
Hyponatremia (Metabolism and nutrition disorders) | 1 (2) | 1 (1) | 3 (3)
Hypophosphatemia (Metabolism and nutrition disorders) | 2 (4) | 1 (5) | 10 (22)
Infections and infestations - Other, specify (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) — Caseating keratin plug with pus on ear drum in R ear removed
Infusion related reaction (General disorders) | 3 (6) | 1 (2) | 20 (57)
Infusion site extravasation (General disorders) | 2 (2) | 0 (0) | 4 (5)
Insomnia (Psychiatric disorders) | 3 (3) | 1 (1) | 10 (10)
Investigations - Other, specify (Investigations) | 1 (1) | 0 (0) | 0 (0) — Low serum iron
Lymphocyte count decreased (Investigations) | 1 (3) | 0 (0) | 0 (0)
Mucositis oral (Gastrointestinal disorders) | 6 (7) | 1 (2) | 22 (38)
Nail loss (Skin and subcutaneous tissue disorders) | 1 (3) | 3 (3) | 10 (10)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 0 (0) | 6 (7)
Neck pain (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0) | 1 (2)
Nervous system disorders - Other, specify (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) — Intermittent imbalance x 1 yr with worsening this pat month
Oral pain (Gastrointestinal disorders) | 4 (4) | 0 (0) | 1 (1)
Pain (General disorders) | 6 (9) | 3 (5) | 30 (59)
Pain in extremity (General disorders) | 5 (6) | 2 (3) | 16 (23)
Palmar-plantar erythrodysesthesia syndrome (Skin and subcutaneous tissue disorders) | 1 (4) | 3 (4) | 7 (9)
Palpitations (Cardiac disorders) | 2 (2) | 0 (0) | 0 (0)
Periodontal disease (Gastrointestinal disorders) | 2 (3) | 0 (0) | 0 (0)
Peripheral sensory neuropathy (Nervous system disorders) | 6 (14) | 3 (5) | 28 (47)
Pharyngeal mucositis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Pharyngolaryngeal pain (General disorders) | 1 (2) | 0 (0) | 0 (0)
Phlebitis (Vascular disorders) | 1 (1) | 0 (0) | 1 (1)
Platelet count decreased (Investigations) | 6 (12) | 0 (0) | 10 (21)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 2 (2)
Postnasal drip (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 3 (3)
Proteinuria (Renal and urinary disorders) | 3 (9) | 0 (0) | 10 (24)
Pruritus (Skin and subcutaneous tissue disorders) | 3 (5) | 2 (2) | 13 (15)
Purpura (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 5 (5)
Rash acneiform (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 2 (4) | 2 (3) | 12 (19)
Sinus tachycardia (Cardiac disorders) | 1 (1) | 0 (0) | 1 (1)
Sinusitis (Infections and infestations) | 3 (4) | 2 (4) | 6 (7)
Skin and subcutaneous tissue disorders - Other, specify (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) — Acquired perforating dermatosis elbows
Skin hyperpigmentation (Skin and subcutaneous tissue disorders) | 1 (1) | 2 (2) | 8 (10)
Skin infection (Infections and infestations) | 5 (5) | 1 (2) | 16 (25)
Skin ulceration (Skin and subcutaneous tissue disorders) | 1 (1) | 2 (2) | 5 (5)
Sore throat (Respiratory, thoracic and mediastinal disorders) | 2 (3) | 0 (0) | 2 (2)
Supraventricular tachycardia (Cardiac disorders) | 1 (2) | 0 (0) | 1 (1)
Thromboembolic event (Vascular disorders) | 1 (1) | 0 (0) | 2 (2)
Toothache (Gastrointestinal disorders) | 2 (2) | 2 (3) | 9 (10)
Upper gastrointestinal hemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Upper respiratory infection (Infections and infestations) | 0 (0) | 2 (3) | 21 (34)
Urinary incontinence (Renal and urinary disorders) | 2 (3) | 0 (0) | 5 (6)
Urinary retention (Renal and urinary disorders) | 1 (3) | 1 (3) | 4 (7)
Urinary tract infection (Infections and infestations) | 2 (2) | 0 (0) | 9 (15)
Urinary tract obstruction (Renal and urinary disorders) | 1 (1) | 0 (0) | 3 (4)
Voice alteration (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 3 (3) | 16 (17)
Vomiting (Gastrointestinal disorders) | 2 (2) | 2 (5) | 9 (15)
Watering eyes (Eye disorders) | 2 (6) | 3 (3) | 27 (27)
Weight loss (Investigations) | 0 (0) | 1 (1) | 19 (39)
White blood cell decreased (Investigations) | 2 (4) | 0 (0) | 1 (1)
Bloating (Gastrointestinal disorders) | 0 (0) | 1 (1) | 1 (1)
Chills (General disorders) | 0 (0) | 2 (3) | 0 (0)
Dry eye (Eye disorders) | 0 (0) | 1 (1) | 2 (3)
Dry mouth (Gastrointestinal disorders) | 0 (0) | 2 (2) | 8 (8)
Dysphagia (Gastrointestinal disorders) | 0 (0) | 1 (2) | 0 (0)
Hemorrhoidal hemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1) | 2 (2)
Hemorrhoids (Gastrointestinal disorders) | 0 (0) | 1 (1) | 5 (5)
Hypomagnesemia (Metabolism and nutrition disorders) | 0 (0) | 2 (7) | 30 (64)
Hypotension (Vascular disorders) | 0 (0) | 1 (2) | 13 (23)
Infections and infestations - Other, specify (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) — Infection with Grade 3 or 4 neutrophils (ANC <1.0 x 10e9/L): Nose
Laryngeal inflammation (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Mucosal infection (Infections and infestations) | 1 (1) | 1 (1) | 0 (0)
Muscle weakness upper limb (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 3 (3) | 2 (3) | 13 (20)
Neutrophil count decreased (Investigations) | 6 (13) | 3 (17) | 26 (68)
Non-cardiac chest pain (Musculoskeletal and connective tissue disorders) | 2 (3) | 1 (1) | 3 (4)
Osteonecrosis of jaw (Musculoskeletal and connective tissue disorders) | 5 (7) | 3 (5) | 13 (19)
Paresthesia (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Pharyngitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Pharyngolaryngeal pain (Gastrointestinal disorders) | 0 (0) | 3 (3) | 0 (0)
Respiratory, thoracic and mediastinal disorders - Other, specify (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) — Rhinorrhea
Skin and subcutaneous tissue disorders - Other, R hallux valgus (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Skin hypopigmentation (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Soft tissue infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Sore throat (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Stomach pain (Gastrointestinal disorders) | 0 (0) | 1 (2) | 0 (0)
Tooth infection (Infections and infestations) | 0 (0) | 1 (1) | 4 (8)
Tremor (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Urinary tract infection (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0)
Vasovagal reaction (Nervous system disorders) | 0 (0) | 1 (1) | 4 (4)
Abdominal distension (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Abdominal infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Alanine aminotransferase increased (Investigations) | 0 (0) | 0 (0) | 6 (8)
Anal hemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Anal ulcer (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Anxiety (Psychiatric disorders) | 0 (0) | 0 (0) | 3 (3)
Arthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Ascites (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Aspartate aminotransferase increased (Investigations) | 0 (0) | 0 (0) | 6 (8)
Atrial fibrillation (Cardiac disorders) | 0 (0) | 0 (0) | 3 (3)
Atrial flutter (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Blood bilirubin increased (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1)
Blurred vision (Eye disorders) | 0 (0) | 0 (0) | 4 (4)
Bronchial infection (Infections and infestations) | 0 (0) | 0 (0) | 6 (8)
Cardiac disorders - Other, L ventricular hypertrophy (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Cataract (Eye disorders) | 0 (0) | 0 (0) | 4 (9)
Cheilitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 5 (5)
Colitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (2)
Conduction disorder (Cardiac disorders) | 0 (0) | 0 (0) | 1 (2)
Conjunctivitis (Eye disorders) | 0 (0) | 0 (0) | 2 (2)
Cytokine release syndrome (Immune system disorders) | 0 (0) | 0 (0) | 1 (1)
Ear and labyrinth disorders - Other, Cerumen impaction b/l-wax removed; (Ear and labyrinth disorders) | 1 (1) | 0 (0) | 1 (1)
External ear inflammation (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 1 (1)
Eye disorders - Other, Blepharitis, R. eye (Eye disorders) | 0 (0) | 0 (0) | 1 (1)
Eye infection (Infections and infestations) | 0 (0) | 0 (0) | 2 (2)
Eye pain (Eye disorders) | 0 (0) | 0 (0) | 2 (2)
Flank pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Flushing (Vascular disorders) | 0 (0) | 0 (0) | 7 (8)
Fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 6 (6)
Gastrointestinal disorders - Other, L arytenoid inflammation (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
General disorders and administration site conditions - Other, specify (General disorders) | 0 (0) | 0 (0) | 1 (1) — Cold intolerance
Glucose intolerance (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (2)
Hallucinations (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1)
Hearing impaired (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 2 (2)
Hematoma (Vascular disorders) | 0 (0) | 0 (0) | 1 (1)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 3 (3)
Hypermagnesemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 3 (3)
Hypokalemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 7 (13)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Injection site reaction (General disorders) | 0 (0) | 0 (0) | 4 (4)
Injury, poisoning and procedural complications - Other, specify (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) — L leg laceration with stitches removed on 9/12/11
Intracranial hemorrhage (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Joint effusion (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Joint range of motion decreased (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 3 (3)
Laryngitis (Infections and infestations) | 0 (0) | 0 (0) | 2 (2)
Lip infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Lower gastrointestinal hemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 2 (2)
Lung infection (Infections and infestations) | 0 (0) | 0 (0) | 6 (7)
Lymphedema (Vascular disorders) | 0 (0) | 0 (0) | 1 (2)
Memory impairment (Nervous system disorders) | 0 (0) | 0 (0) | 2 (2)
Muscle weakness lower limb (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 6 (9)
Muscle weakness trunk (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Musculoskeletal and connective tissue disorder - Other, specify (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) — Compression fracture
Nail discoloration (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 10 (10)
Nail infection (Infections and infestations) | 0 (0) | 0 (0) | 4 (4)
Nail ridging (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 3 (3)
Nausea (Gastrointestinal disorders) | 4 (4) | 2 (4) | 16 (22)
Nervous system disorders - Other, specify (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) — Dystonic reaction
Optic nerve disorder (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 1 (1)
Oral dysesthesia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Otitis externa (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 1 (1)
Otitis media (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 1 (1)
Pain of skin (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Peripheral motor neuropathy (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Personality change (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1)
Pharyngolaryngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 5 (5)
Productive cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 4 (4)
Rectal fistula (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Rectal hemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 10 (13)
Rectal pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 3 (6)
Renal and urinary disorders - Other, Acute R hydronephrosis (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1)
Respiratory, thoracic and mediastinal disorders - Other, specify (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 13 (13)
Salivary gland infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Scrotal pain (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 1 (1)
Sinus bradycardia (Cardiac disorders) | 0 (0) | 0 (0) | 2 (2)
Sinus disorder (Cardiac disorders) | 0 (0) | 0 (0) | 2 (2)
Skin and subcutaneous tissue disorders - Other, Actinic Keratosis (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Skin atrophy (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Skin induration (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 2 (2)
Suicidal ideation (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1)
Syncope (Nervous system disorders) | 0 (0) | 0 (0) | 4 (4)
Transient ischemic attacks (Cardiac disorders) | 0 (0) | 0 (0) | 2 (2)
Upper respiratory infection (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 21 (34)
Urinary frequency (Renal and urinary disorders) | 0 (0) | 0 (0) | 2 (3)
Urinary tract pain (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1)
Urticaria (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Vascular disorders - Other, Conjunctival hemorrhage b/l (Vascular disorders) | 0 (0) | 0 (0) | 1 (1)
Ventricular arrhythmia (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Wheezing (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Wound infection (Infections and infestations) | 0 (0) | 0 (0) | 4 (4)
Skin and subcutaneous tissue disorders - Other, angiomas (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Skin and subcutaneous tissue disorders - Other, chrondrodermatitis nodularis helicus (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Skin and subcutaneous tissue disorders - Other, Corn-like lesion R heel (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Skin and subcutaneous tissue disorders - Other, Depession L temporal area (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Skin and subcutaneous tissue disorders - Other, Erythema (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Skin and subcutaneous tissue disorders - Other, Ingrown toenail, medial R big toe (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Skin and subcutaneous tissue disorders - Other, L foot halux bunion (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Skin and subcutaneous tissue disorders - Other, nail splinter hemorrhages (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Skin and subcutaneous tissue disorders - Other, skin breakdown on R hip (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Skin and subcutaneous tissue disorders - Other, skin fragility and thinning (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Skin and subcutaneous tissue disorders - Other, symptomatic corn on R lateral foot (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Ear and labyrinth disorders - Other, Cerumen impaction, b/l (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 1 (1)
Ear and labyrinth disorders - Other, Ear discharge (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 1 (1)
Ear and labyrinth disorders - Other, Perforated ear drum (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 1 (1)
Gastrointestinal disorders - Other, Loss of crown to dental implant #14 (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Gastrointestinal disorders - Other, Cracked tooth (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Gastrointestinal disorders - Other, Fracture tooth #14 (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Gastrointestinal disorders - Other, Gingival bleeding (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Gastorintestinal disorders - Other, Gum swelling (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (2)
Gastrointestinal disorders - Other, Gum swelling, intermittent (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Infections and infestations - Other, Jaw infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Infections and infestations - Other, R jaw infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Infections and infestations - Other, Viral (Infections and infestations) | 1 (1) | 1 (1) | 0 (0)
Infections and infestations - Other, Specify (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) — Infection with normal ANC or Grade 1 or 2 neutrophils:Stomach
Infections and infestations - Other, Strep throat diagnosed at Kaiser (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Infections and infestations - Other, upper eye lid - chalazion (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Infections and infestations - Other, Fungal:oral candidiasis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Infections and infestations - Other, Specify (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) — Gastrointestinal-Aeromonas Veronii
Infections and infestations - Other, Oral fungal (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Infections and infestations - Other, Stool (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Infections and infestations - Other, Specify (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) — Subgingival, R mandible suggestive of ONJ
Skin and subcutaneous tissue disorders - Other, Bruising and fragility of skin (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Skin and subcutaneous tissue disorders - Other, Eschar on L. buttock (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Skin and subcutaneous tissue disorders - Other, Specify (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) — Poor wound healing at extraction site of tooth #31
Renal and urinary disorders - Other, Bleeding at nephrostomy tube site (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1)
Renal and urinary disorders - Other, CR CL < 50 (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1)
Renal and urinary disorders - Other, Decreased urinary flow (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1)
Renal and urinary disorders - Other, R hydronephrosis (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1)
Renal and urinary disorders - Other, Urinary hesitancy (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1)
Vascular disorders - Other, L ear bleeding (Vascular disorders) | 0 (0) | 0 (0) | 1 (1)
Vascular disorders - Other, Raynaud Syndrome symptoms (Vascular disorders) | 0 (0) | 0 (0) | 1 (1)
Musculoskeletal and connective tissue disorders - Other, Specify (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) — Muscle cramps/myalgia grade change over baseline
Musculoskeletal and connective tissue disorders, Other, R ankle sprain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Eye disorders - Other, Erythema b/l eyes (Eye disorders) | 0 (0) | 0 (0) | 1 (1)
Eye disorders - Other, Eye cyst (Eye disorders) | 0 (0) | 0 (0) | 1 (1)
Eye disorders - Other, Visual changes, intermittent (Eye disorders) | 0 (0) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2017-01-12): https://cdn.clinicaltrials.gov/large-docs/78/NCT00942578/Prot_SAP_ICF_000.pdf